CLINICAL TRIAL: NCT01620021
Title: Feasibility of Wearable Sensors to Determine Gait Parameters
Status: Completed | Type: Observational
Sponsor: University of South Florida (Other)
Responsible Party: Principal Investigator, Stephanie L. Carey, Assistant Research Professor, University of South Florida
Other Study IDs: Pro00003205
Record Dates: First submitted 2012-06-12; First posted 2012-06-15 (Estimated); Last update posted 2015-05-07 (Estimated); Status verified 2015-05

CONDITIONS: Gait Analysis
Keywords: wearable sensors; kinematics; gait

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Healthy: Ten healthy volunteers with no history of gait and balance issues will be recruited to participate in the study.The participants must be between 18 and 65 years of age.

SUMMARY:
Hypotheses:

• A wearable sensor system can be used to accurately monitor three common gait parameters: gait speed, stride length, and torso motion.

Objectives:

This study will examine the feasibility of using wearable sensors to monitor common gait parameters: gait speed, stride length and torso motion. A wearable sensor system of 8 commercially available inertial measurement units (IMU) will be composed. These sensors will work in unison to monitor the gait parameters.

Technical Objectives

* Gather information on commercially available IMUs
* Use computer software to monitor and record data from IMUs
* Develop an algorithm that can monitor volunteer gait speed, stride length and torso motion
* Develop a graphical algorithm that compares healthy patient data to potential mild traumatic brain injury (mTBI ) candidates
* Determine if there is a potential for mTBI determination using the wearable sensors
* Accurately validate the wearable sensor system to the gait parameters measured using a Vicon motion analysis system

DETAILED DESCRIPTION:
This study will examine the feasibility of using wearable sensors to monitor common gait parameters. A sensor system consisting of 8 wearable inertial measurement units (IMU) that include accelerometers, gyroscopes and magnetometers will be examined. These sensors will be programmed to work in unison to monitor gait parameters. The wearable sensor suite will have the capability to collect and store gait parameter data. The size and weight of each sensor should be similar to a standard metal wrist watch. The sensor suite will monitor three gait parameters: gait speed, stride length, and torso motion. These gait parameters are important for monitoring and detection of mild traumatic brain injury and as well as other neurological and vestibular disorders.

The wearable sensor suite will have the following design parameters:

* Devices must be able to both stream data real-time and record data onboard for later transfer to a computer.
* Data must be processed using a software analysis package such as MATLAB®
* Device must be no heavier than the size of a metal wrist watch
* Device must be easily put on and be easily operated by clinicians and users
* Device must have a battery life of greater than 4 hours The wearable sensor suite will then be validated using an eight camera Vicon infrared optical capture motion analysis system for comparison. Ten healthy volunteers will be asked to complete four different types of gait trials 5 times for each trial type while being monitored by the Vicon motion analysis system and the wearable sensor system.

The types of gait trials will be the following:

* Walk down a 20 ft path at self-selected normal stride length and cadence
* Walk down a 20 ft path with increased stride length while decreasing gait speed
* Walk down a 20 ft path with increased stride length while increasing gait speed
* Walk down a 20 ft path with decreased stride length while decreasing gait speed
* Walk down a 20 ft path with decreased stride length while increasing gait speed

ELIGIBILITY:
Inclusion Criteria:

* no history of gait and balance issues
* 18-65

Exclusion Criteria:

* younger than 18
* older than 65
* problems with gait and balance

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Ten healthy volunteers with no history of gait and balance issues will be recruited to participate in the study. The participants must be between 18 and 65 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2011-04; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
gait speed | 60 seconds
stride length | 60 seconds
Torso motion | 60 seconds
Head motion | 60 seconds

CONTACTS AND LOCATIONS:
Locations (1):
- University of South Florida Motion Analysis Laboratory, Tampa, Florida, United States